CLINICAL TRIAL: NCT06554418
Title: What Works to Prevent Violence Against Women and Girls: Evaluation of the Communities Care Program in Somalia
Brief Title: What Works to Prevent Violence Against Women and Girls in Somalia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Comitato Internazionale per los Sviluppo dei Popoli (CISP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00418976
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Violence Prevention

STUDY DESIGN:
Intervention Model Description: Randomized at the districts level in two regions of Somalia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communities Care (Experimental): Districts in two regions of Somalia randomized to Communities Care violence prevention program with adults and adolescents
  Interventions: Behavioral: Communities Care
- Control (No Intervention): Districts in two regions of Somalia randomized to control - usual programming related to prevention of violence

INTERVENTIONS:
Behavioral: Communities Care — Communities Care is a violence prevention program targeting social norms and behavioral change
  Arms: Communities Care

SUMMARY:
The Communities Care (CC) program has demonstrated promise in changing harmful social norms associated with Gender-based violence (GBV) and increasing confidence in services for women and girls. Therefore, the study will adapt the existing CC program based on previous learnings with adults and expand programming to include adolescent boys and girls, creating the CC adult and CC adolescent program. The CC program intervention implementation will be led by Comitato Internazionale per lo Sviluppo dei Popoli (CISP) non-Governmental Organization (NGO) in partnership with Somalia Ministry of Education and local Women led Organizations (WLO), public schools and mapped GBV and child protection (CP) service providers in Banadir and Galmudug regions of Somalia.

Johns Hopkins will collaborate with local research colleagues to evaluate the CC adult and CC adolescent program. The study will use a hybrid type 2 effectiveness-implementation design guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework. Quantitative methods will be used to measure outcomes at baseline and endline (24 months post baseline) with adults and adolescents (10 and older) participants in the CC programs in intervention compared to control districts in the two regions (Banadir and Galmudug) in South Central Somalia. Quantitative methods will also be used to measure outcomes with adults and adolescents (10 years and older) community members (members that do not participate in the CC program) in intervention and control districts in the 2 regions at baseline, midline (12-months), endline (24-months) and maintenance (36 months). In addition, quantitative and qualitative methods at midline and endline will be used to measure the CC adult and CC adolescent intervention reach, adoption, implementation and maintenance in intervention districts in the two regions.

DETAILED DESCRIPTION:
What Works to Prevent Violence Against Women and Children (FCDO funded) has funded a collaboration between Johns Hopkins and Comitato Internazionale per lo Sviluppo dei Popoli (CISP) NGO in partnership with Somalia Ministry of Education and local researchers and Women led Organizations (WLO) to evaluate the Communities Care (CC) violence prevention intervention with both adults and adolescent in community and school-based settings in two regions of Somalia. The study will use a hybrid type 2 effectiveness-implementation design guided by the RE-AIM framework (e.g., reach, effectiveness, adoption, implementation and maintenance). Quantitative methods will be used to measure violence, health and social norms outcomes with adults (18 and older) and adolescents (10 and older) with participants in CC intervention districts and control districts in the two regions (Banadir and Galmudug) in South Central Somalia. Quantitative methods will also be used to measure outcomes with adults and adolescents (10 years and older) community members (members that do not participate in the CC program) in intervention and control districts in the 2 regions at baseline, midline (12-months), endline (24-months) and maintenance (36 months). In addition, quantitative and qualitative methods at midline and endline will be used to measure the CC adult and CC adolescent intervention reach, adoption, implementation and maintenance in intervention districts in the two regions.

ELIGIBILITY:
Inclusion Criteria

* Age 10 years or older
* Participant in CC adult or CC adolescent program in collaboration with 9 public schools in districts randomized to intervention or control in two regions of Somalia
* Living/resident of target districts (including internally displaced persons (IDPs) and does not have plans to move/leave the district or surrounding area in the next 12 months (this is critical for the longitudinal data collection with CC program participants)

Exclusion Criteria:

* Less than 10 years old
* Not a participant in CC adult or CC adolescent
* Not a resident of target districts-

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — self-identified as male and female adolescents and adults
Enrollment: 3500 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Cyber-Sexual Harassment survey score | 9 and 12 months
  Adolescent report of experience of peer-to-peer or adult on-line and in-person harassment, Mean scale score ranges from 1 to 5 with higher scores being worse outcome
Peer-to-peer physical and sexual violence in school and community survey score | 9 and 12 months
  Adolescent report of experience of peer to peer violence in schools, Mean scale score ranges from 1 to 5 with higher scores being worse outcome
Harsh punishment in school as assessed by the Parent-Child Conflict Scale adapted for teachers | 9 and 12 months
  Adolescent report of witness or experience harsh punishment in school using the Parent-Child Conflict Tactics Scale adapted for teachers, Mean scale score 1-5, with higher score being worse outcome
Witnessing intimate partner violence (IPV) survey score | 9 and 12 months
  Adolescent report of witnessing IPV in the household, mean scale score ranges from 1 to 5 with higher scores being worse outcome
Harsh Punishment in Household as assessed by the Parent-Child Conflict Scale | 9 and 12 months
  Adolescent report of witness and experience harsh punishment in household using Parent-Child Conflict Tactics Scale, mean scale score ranges from 1 to 5 with higher scores being worse outcome
IPV victimization and/or perpetration as assessed by Somalia National Survey | 9 and 12 months
  Adult report of experience and/or perpetration of IPV, mean scale score ranges from 1 to 5 with higher scores being worse outcome
Use of Harsh Punishment in Household as assessed by the Parent-Child Conflict Tactics Scale | 9 and 12 months
  Adult report of use of harsh punishment, mean scale score ranges from 1 to 5 with higher scores being worse outcome
Non-partner harassment as assessed by the National Somalia Survey | 9 and 12 months
  Adult report of non-partner harassment, mean scale score ranges from 1 to 5 with higher scores being worse outcome
Non-partner physical and/or sexual violence victimization as assessed by the National Somalia Survey | 9 and 12 months
  Adult report of physical and/or sexual violence victimization by non-partner, mean scale score ranges from 1 to 5 with higher scores being worse outcome

SECONDARY OUTCOMES:
Personal Beliefs and Social Norms about Gender Based Violence as assessed by the Social Norms and Beliefs about Gender Based Violence Scale | 9 and 12 months
  Adolescent and adult personal beliefs and social norms about gender based violence, mean scale scores range from 1-5, higher scores being worse outcome
Gender equality survey score | 9 and 12 months
  Adult and adolescent report of equality in access to education, resources and decision making between women/girls and men/boys, mean scale score range from 1-5, higher score is worse outcome
IPV acceptability survey score | 9 and 12 months
  Adult and adolescent report on acceptability of intimate partner violence (IPV), for example, It is justifiable for a husband to hit his wife because she argues with him, it is acceptable for a husband to force his wife to have sex when she does not want to. mean subscale score range from 1-5, higher score is worse outcome
Sexual and reproductive health knowledge and empowerment score | 9 and 12 months
  Adolescent knowledge in the domains of puberty, female genital mutilation (FGM), child marriage, and sexually transmitted infection (STI) and empowerment measured for puberty, child marriage, FGM, PV, and contraception use, mean scale score range from 1-5, higher score is better outcomes
Confidence in service providers (adolescents and adults) score | 9 and 12 months
  Adolescent and adult report on confidence in service providers in responding to gender based violence across several sectors (health care, justice system, elders, psychosocial services and community health workers). Mean scale score range from 1-5, higher score is better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Glass, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- CISP Somalia, Mogadishu, Wadajir District, Somalia